CLINICAL TRIAL: NCT02466282
Title: A Randomized Controlled Comparison of Optical Coherence Tomography Guidance and Angiography-only Guidance for Percutaneous Coronary Intervention With Bioresorbable Vascular Scaffold
Brief Title: A Comparison of Optical Coherence Tomography Guidance and Angiography-only Guidance for Percutaneous Coronary Intervention With Bioresorbable Vascular Scaffold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2015-0019
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Angiography-guidance (Active Comparator): Everolimus-eluting bioresorbable vascular scaffold (Absorb, Abbott Vascular, Santa Clara, CA, USA) was made from a bioabsorbable polylactic acid backbone which is coated with a more rapidly absorbed polylactic acid layer that contains and controls the release of the antiproliferative drug, everolimus. PCI will be performed with BVS under conventional coronary angiography without any other intravascular imaging modality.
  Interventions: Device: Angiography-guided PCI with bioresorbable vascular scaffold
- OCT-guidance (Experimental): Everolimus-eluting bioresorbable vascular scaffold (Absorb, Abbott Vascular, Santa Clara, CA, USA) was made from a bioabsorbable polylactic acid backbone which is coated with a more rapidly absorbed polylactic acid layer that contains and controls the release of the antiproliferative drug, everolimus. For optimized PCI, both conventional coronary angiography and optical coherence tomography can be used before and after stent implantation. OCT study should be checked at the final post-procedure and stent implantation is optimized.
  Interventions: Device: optical coherence tomography-guided PCI with bioresorbable vascular scaffold

INTERVENTIONS:
Device: Angiography-guided PCI with bioresorbable vascular scaffold — Everolimus-eluting bioresorbable vascular scaffold (Absorb, Abbott Vascular, Santa Clara, CA, USA) was made from a bioabsorbable polylactic acid backbone which is coated with a more rapidly absorbed polylactic acid layer that contains and controls the release of the antiproliferative drug, everolimus. PCI will be performed with BVS under conventional coronary angiography without any other intravascular imaging modality.
  Arms: Angiography-guidance
Device: optical coherence tomography-guided PCI with bioresorbable vascular scaffold — Everolimus-eluting bioresorbable vascular scaffold (Absorb, Abbott Vascular, Santa Clara, CA, USA) was made from a bioabsorbable polylactic acid backbone which is coated with a more rapidly absorbed polylactic acid layer that contains and controls the release of the antiproliferative drug, everolimus. For optimized PCI, both conventional coronary angiography and optical coherence tomography can be used before and after stent implantation. OCT study should be checked at the final post-procedure and stent implantation is optimized.
  Arms: OCT-guidance

SUMMARY:
It is well-known that non-optimal stent implantation associated with under-expansion or incomplete strut apposition during percutaneous coronary intervention (PCI) leads to a higher incidence of restenosis and stent thrombosis. OCT-guided PCI with metallic stent has previously been shown to be safe and feasible, resulting in better clinical outcomes compared with angiography-only guided PCI. Everolimus-eluting bioabsorbable vascular scaffold (BVS; Abbott Vascular, Santa Clara, CA, USA) was made from a bioabsorbable polylactic acid backbone which is coated with a more rapidly absorbed polylactic acid layer that contains and controls the release of the antiproliferative drug, everolimus. BVS has a number of proposed advantages over current metallic stent technology. These include elimination of chronic sources of vessel irritation and inflammation, which can reduce the potential risk of late scaffold thrombosis after complete scaffold bioresorption. Although the current generation of the Absorb BVS have larger strut thickness of 150 μm compared with 80 μm of strut of Xience stent, the acute recoil of the polymeric device was similar to that of metallic stent. However, operators tented to use dilating devices less aggressively because of the concerns about limitation in elongation-at-break of polylactide. Previous studies reported 20-30% of under-expansion or malapposition with BVS, which would increase the risk of adverse events including late stent thrombosis. OCT-guidance may improve more optimized scaffold placement and also better outcomes. Therefore, investigators will compare OCT guidance and angiography-only guidance for PCI with BVS regarding incomplete scaffold apposition and neointimal scaffold coverage. Investigators are also going to compare these two strategies regarding clinical outcomes with verification of the cut-off value by OCT-acquired uncovered scaffold rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old
* Patients with ischemic heart disease who are considered for coronary revascularization with PCI
* Significant coronary de novo lesion (stenosis > 70% by quantitative angiographic analysis) treated by single BVS ≤ 25mm
* Reference vessel diameter of 2.5 to 3.5 mm by operator assessment

Exclusion Criteria:

* Myocardial infarction
* Complex lesion morphologies such as aorta-ostial, unprotected left main, chronic total occlusion, graft, thrombosis, and restenosis
* Reference vessel diameter <2.5 mm or >3.5 mm
* Heavy calcified lesions (definite calcified lesions on angiogram)
* Lesions requiring 2 or more BVS
* Contraindication or hypersensitivity to anti-platelet agents or contrast media
* Treated with any metallic stent or BVS within 3 months at other vessel
* Creatinine level ≥ 2.0 mg/dL or ESRD
* Severe hepatic dysfunction (3 times normal reference values)
* Pregnant women or women with potential childbearing
* Inability to follow the patient over the period of 1 year after enrollment, as assessed by the investigator
* Inability to understand or read the informed content

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Percentage of uncovered scaffold struts | six months
  Percentage of uncovered scaffold struts between OCT guidance vs. angiography-only guidance PCI on 6 month OCT

SECONDARY OUTCOMES:
Major cardiac and cerebrovascular adverse events (MACCEs) | until one year
  Cardiac death, myocardial infarction, target vessel revascularization, stent thrombosis, cerebrovascular accident and major bleeding between OCT guidance vs. angiography-only guidance PCI until 12 months
  *Major bleeding ; causing mortality, hypovolemic shock or severe hypotension requiring inotropes or surgery, intrapericardial with tamponade, significant disabling (e.g. intraocular bleeding leading to loss of vision), symptomatic intracranial haemorrhage, intraocular bleeding leading to loss of vision, hemoglobin drop ≥ 3g/dL, or requiring transfusion more than 2 units
Percentage of incomplete scaffold struts apposition | six months after stent implantation
  Scaffold strut malapposition: Malapposition is defined by a clear seperation between the abluminal side of the strut and the vessel wall. As a result, scaffold malapposition is defined as the presence of any malapposed struts. percentage of malapposed struts (% malapposed strut) was the ratio of malapposed struts from total analyzable struts.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea